CLINICAL TRIAL: NCT05692297
Title: Denosumab Treatment in Patients With Chronic Kidney Disease (CKD) at High Risk of Fracture: A Prospective, Randomised Controlled Study
Brief Title: Denosumab Treatment in CKD Patients at High Risk of Fracture
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Capital Medical University (Other)
Responsible Party: Principal Investigator, Dongliang Zhang, MD, Director of Nephrology Department of Beijing Jishuitan Hospital, Capital Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: K2022-203-00
Record Dates: First submitted 2023-01-11; First posted 2023-01-20 (Actual); Last update posted 2023-01-25 (Actual); Status verified 2023-01

CONDITIONS: Chronic Kidney Diseases; Fracture; Bone Density, Low; End Stage Renal Disease
Keywords: Denosumab; Chronic Kidney Diseases; Treatment; Fracture
MeSH Terms: conditions — Renal Insufficiency, Chronic; Fractures, Bone; Bone Diseases, Metabolic; Kidney Failure, Chronic | interventions — Denosumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Denosumab group (Experimental): Fifty-one patients were randomly assigned to the denosumab group, which received subcutaneous injection of denosumab 60mg once every 6 months. Serum calcium, phosphorus, alkaline phosphatase, iPTH, tPINP, 25(OH)VitD, DXA and qCT were measured before medication. Serum calcium, phosphorus and iPTH were examined at day 1, 7 and 14, alkaline phosphatase, tPINP and 25(OH)VitD at day 7 and 14, and electrocardiogram at day 1 and 7 after treatment. Intravenous calcium supplementation was required if muscle spasms and QT prolongation occurred. Six months after medication, subcutaneous injections of denosumab 60mg were repeated. The protocol was repeated every 6 months, totally 24 months. Bone mineral density, clinical parameters and adverse events were evaluated at 24 months.
  Interventions: Drug: Denosumab
- Non-denosumab group (Active Comparator): The other 51 patients did not use denosumab and used other medications, such as diphosphonates, active vitamin D and/or active vitamin D analogue, calcimimetics, calcitonin, estrogen receptor agonists, etc. At the same time, calcium and vitamin D were supplemented. The baseline serum calcium, phosphorus, alkaline phosphatase, iPTH, tPINP, 25(OH)VitD, DXA, and qCT were measured. The above parameters were rechecked every 6 months, and the medications was recorded, totally 24 months.
  Interventions: Drug: Non-denosumab

INTERVENTIONS:
Drug: Denosumab — The patients in the denosumab group received subcutaneous injection of denosumab 60mg once every 6 months for 24 months.
  Arms: Denosumab group
Drug: Non-denosumab — Taken other medications, such as diphosphonates, active vitamin D and/or active vitamin D analogue, calcimimetics, calcitonin, estrogen receptor agonists, etc.
  Arms: Non-denosumab group

SUMMARY:
Objective: To verify the efficacy and safety of denosumab in the prevention and treatment of CKD-MBD in CKD patients with high risk of fracture.

Methods: A cohort of CKD patients with high risk of fracture was established and followed up for long periods (≥24 months). Patients with CKD3b-5D stage and fracture risk assessment tool (FRAX) scores at high risk or very high risk of fracture were enrolled. A multicenter, prospective, open-label, randomised controlled, interventional study was conducted. The patients were divided into two groups. The patients in the denosumab group received subcutaneous injection of denosumab 60mg once every 6 months, and the patients in the non-denosumab group received conventional treatment. Bone metabolic markers (serum calcium, phosphorus, vitamin D, parathyroid hormone, alkaline phosphatase, tartrate-resistant acid phosphatase 5b, osteocalcin, total N-terminal propeptide of type I collagen, etc.), bone mineral density (dual-energy X-ray, quantitative CT), and vascular calcification score were regularly monitored. All adverse events (all-cause death, cardiovascular death, cardiac events, fracture, hospitalization, emergency department visits, etc.) were recorded during the follow-up period. Bone mineral density and clinical parameters were compared between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years old;
* Stage 3b-5D chronic kidney disease;
* The 10-year probability of hip fracture assessed by fracture risk assessment tool (FRAX) was >5%;
* Voluntarily signed informed consent.

Exclusion Criteria:

* Age < 18 or ≥100 years;
* Premenopausal women;
* Denosumab was absolutely contraindicated;
* Had received denosumab or bisphosphonates therapy;
* Tertiary hyperparathyroidism;
* Patients with malignant tumor;
* Patients at risk for osteonecrosis of the jaw;
* Estimated follow-up time ≤12 months.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of bone mineral density (BMD) decline at the lumbar spine | 24 months
  Rate of BMD decline =[(BMD24-BMD Baseline)÷BMD baseline]*100%

SECONDARY OUTCOMES:
Rate of fresh fractures, cardiovascular cerebrovascular adverse events and all-cause mortality | 24 months
  Fresh fractures were new non-traumatic fractures during follow-up. Cardiovascular cerebrovascular adverse events were Acute myocardial infarction, heart failure, shock, cardiac arrest, stroke, and lower limb arterial occlusion occurred during follow-up. All-cause mortality was death from any cause during follow-up.

CONTACTS AND LOCATIONS:
Locations (1):
- Nephrology Department of Beijing Jishuitan Hospital, Beijing, Beijing Municipality, China